CLINICAL TRIAL: NCT06196242
Title: Research on Lead Localization for Deep Brain Stimulation After Implantation
Brief Title: Deep Brain Stimulation Lead Localization After Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Luming Li, Professor, Tsinghua University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LeadLocMRI
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Lead Localization; MRI
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBS lead localization (Experimental): Participates will receive a head MRI anc CT scan. The stimulation target and the related neural nuclei will be reconstructed using MRI images. The spatial position of the implanted lead will be identified with MRI and CT. Through comparing with the identified lead position by CT, the accuracy of lead localization by MRI will be evaluated.
  Interventions: Diagnostic Test: MRI and CT scan

INTERVENTIONS:
Diagnostic Test: MRI and CT scan — An MRI scan of the head in about 30 minutes. During the scan, MRI thermometry will be performed to monitor for possible lead heating due to the interaction of the MRI radiofrequency field and the implanted devices.
  An CT plain scan of the head in about 10 minutes.

SUMMARY:
Deep brain stimulation (DBS) is an effective treatment for a variety of neurological and psychiatric disorders, with more than 200,000 patients implanted with DBS devices worldwide. Parkinson's disease is one of the typical indications.The clinical outcomes of DBS depends on the accurate implantation of the lead, and the identification of the lead locations is the basis for evaluating the effectiveness of the treatment. The aim of this study is to localize the implantation position of the lead based on postoperative MRI images and to reconstruct the relative spatial relationship between the lead and the stimulation target. By comparing with the lead position identified based on postoperative CT, this study will evaluate the accuracy of identifying the DBS lead position directly from MRI. This study may help to optimise the stimulation parameters and investigate the best stimulation targets for DBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients with DBS devices, DBS implanted for at least 1 month.
* Ability to tolerate DBS turn-off for at least 30 minutes.
* DBS devices do not contain the ferromagnetic material.
* The patients can fully understand the content of the trial and sign the informed consent form.
* Able to comply to the requirements of this study.

Exclusion Criteria:

* Presence of other concomitant diseases that have or require implantation of pacemakers, defibrillators, cochlear implants, or other neurostimulation devices.
* Patients who are abnormally sensitive to temperature or allergic to heat.
* Patients with severe psychiatric disorders or cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Lead position | 1 day
  The accuracy of the lead localization will be evaluated by the distance between the identified position of the lead electrode and the center of the reconstructed stimulation target. The result of lead localization by CT will be used as the reference.

CONTACTS AND LOCATIONS:
Locations (1):
- National Engineering Research Center of Neuromodulation, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No